CLINICAL TRIAL: NCT06158607
Title: Development and Pilot Testing of an Addiction Clinic-Based PrEP Adherence Intervention for Women with Substance Use Disorders
Brief Title: Pre-exposure Prophylaxis (PrEP) Adherence Intervention for Women with Substance Use Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Angela M Heads, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-21-0451
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Substance Use
Keywords: Pre-Exposure Prophylaxis; Women; HIV Prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Addiction Clinic-Based PrEP Adherence Intervention for Women with Substance Use Disorders
- Standard of care treatment (Active Comparator)
  Interventions: Other: Standard of care treatment

INTERVENTIONS:
Behavioral: Addiction Clinic-Based PrEP Adherence Intervention for Women with Substance Use Disorders — Provision of PrEP information through 4 counseling sessions, prevention navigation, and nurse practitioner prescribed PrEP in an addiction treatment setting.
  Arms: Intervention
Other: Standard of care treatment — Participants in substance use treatment will be given information and referral to a community partner who will evaluate them to determine if they could benefit from PrEP for HIV prevention
  Arms: Standard of care treatment

SUMMARY:
The goal of this clinical trial is to test an addiction-clinic based behavioral intervention for increasing PrEP uptake and adherence among women who engage in high-risk sexual behaviors and problematic substance use. The main question it aims to answer is:

• If the integrated intervention increase PrEP uptake and adherence compared to standard treatment

Participants will

* receive provision of PrEP information through 4 counseling sessions
* prevention navigation
* receive nurse practitioner prescribed PrEP in an addiction treatment setting

Researchers will compare intervention group with standard treatment to see if the integrated intervention help increase PrEP uptake and adherence

ELIGIBILITY:
Inclusion Criteria:

* Black/African American and Hispanic/Latina cisgender women
* diagnosed with a Substance use disorder (SUD) per Diagnostic and Statistical Manual of Mental Illnesses (DSM)-5 criteria
* HIV negative
* sexually active with an opposite sex partner within the past 6 months
* not using PrEP for HIV prevention at the time of screening
* able to speak, read, and write in English; and
* own or have regular access to a smart phone.

Exclusion Criteria:

* be concurrently participating in another SUD behavioral treatment program
* unable to provide informed consent for participation (e.g., have severe cognitive impairment that would interfere with their ability to consent, understand study procedures and/or effectively participate in therapy
* have psychological distress that would prohibit them from participating in the study
* be unable or unwilling to meet study requirements
* be ineligible for PrEP based on Centers for Disease Control and Prevention (CDC)-defined criteria for PrEP based on substance use and sexual risk
* have medical contraindications for PrEP (e.g., known renal impairment which can be exacerbated by PrEP use).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake | 12 weeks post intervention
  Filling the PrEP prescription and taking at least one dose of the medication by two weeks following their visit with the PrEP provider

SECONDARY OUTCOMES:
Daily PrEP adherence as assessed by the levels of tenofovir (TFV) urine concentrations | 90 days post PrEP initiation
  levels of tenofovir (TFV) urine concentrations (>1000ng/ml) detected in urine shows higher adherence
Daily PrEP adherence as assessed by the proportion of videos uploaded | 12 weeks post PrEP initiation
Daily PrEP adherence as assessed by the proportion of self reported daily adherence | 12 weeks post PrEP initiation
Enrollment rate as assessed by the number of participants that signed the consent form | 12 weeks post intervention
Number of sessions attended by participants | 12 weeks post enrollment
Study retention as assessed by the number of participants that completed the study | 12 weeks post enrollment
Intervention acceptability as assessed by the Client satisfaction questionnaire | 12 weeks post intervention
  This is a 15 item questionnaire and each is cored from 1(not at all true)-9( absolutely true), higher number indicating more satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Angela Heads, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Louis A. Faillace, MD, Department of Psychiatry and Behavioral Sciences, University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heads AM, Santa Maria D, Hill MJ, Suchting R, Evans KN, Gaul Z, Yammine L, de Dios C, Schmitz JM. Development and Pilot Testing of an Addiction Clinic-Based Pre-Exposure Prophylaxis Uptake and Adherence Intervention for Women with Substance Use Disorders: Protocol for a Pilot Randomized Trial. JMIR Res Protoc. 2025 May 23;14:e64961. doi: 10.2196/64961. PMID 40409752